CLINICAL TRIAL: NCT05102656
Title: Patient Perceptions of the Relational Empathy of Healthcare Practitioners From the Department of Emergency Medicine During COVID-19: A Randomized, Controlled Trial Comparing In-Person Interaction With Personal Protective Equipment (PPE) Versus Video Interaction Without PPE
Brief Title: Patient Perceptions of the Relational Empathy of Healthcare Practitioners From the Department of Emergency Medicine During the COVID-19 Pandemic
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2020-1298; NCI-2021-10960 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-1298 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-10-29; First posted 2021-11-01 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: COVID-19 Infection; Hematopoietic and Lymphoid Cell Neoplasm; Malignant Solid Neoplasm
MeSH Terms: conditions — COVID-19; Hematologic Neoplasms | interventions — Practice Guidelines as Topic; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (video call) (Other): Patients receive standard of care via video call with treating physician.
  Interventions: Procedure: Discussion; Other: Questionnaire Administration
- Group B (in-person) (Other): Patients receive standard of care in-person physician visits.
  Interventions: Other: Best Practice; Other: Questionnaire Administration

INTERVENTIONS:
Other: Best Practice — Physician conversations occur in-person
  Other Names: standard of care; standard therapy
  Arms: Group B (in-person)
Procedure: Discussion — Physician conversations occur via video call
  Other Names: Discuss
  Arms: Group A (video call)
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This study investigates patients' perceptions of their doctor's or nurse's empathy during an in-person interaction with the doctor or nurse wearing personal protective equipment (PPE) compared to during a video interaction with the doctor or nurse without PPE. The goal of this research study is to learn whether patients who visit the Acute Cancer Care Center at MD Anderson believe they get better (more empathetic) care from doctors who visit them in person wearing PPE or from doctors who visit them by video call and do not wear PPE.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine whether patients perceive their healthcare practitioner as more empathetic during an in-person interaction with the practitioner wearing personal protective equipment (PPE), or during a video interaction without the need for PPE.

SECONDARY OBJECTIVES:

I. To assess whether certain physicians perform better with video whereas others perform better in person.

II. To characterize generational differences in patient perception of healthcare practitioner empathy during an in person interaction with the practitioner wearing PPE, or during a video interaction without the need for PPE.

OUTLINE: After initial visit, patients are randomized to 1 of 2 groups.

GROUP A (NO PPE): Patients receive standard of care via video call with treating physician.

GROUP B (WEARING PPE): Patients receive standard of care in-person physician visits.

ELIGIBILITY:
Inclusion Criteria:

* >= 18 years old
* Able to speak and write in English
* Able to understand and willing to sign a written informed consent document
* Willing and able to complete the study assessment(s)

Exclusion Criteria:

* Refuses to participate
* Too ill to participate, in the estimation of the patient's physician

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2021-06-02 (Actual); Primary Completion 2027-02-02 (Estimated); Study Completion 2027-02-02 (Estimated)

PRIMARY OUTCOMES:
Patients' perceptions of healthcare provider empathy | Through study completion, an average of 1 year
  Univariate linear regression analysis will be used to determine the association between the approach (in-person interaction/with personal protective equipment [PPE] versus video interaction/without PPE) and the composite scores or scores for each question (for each of the two tools [the CARE Measure and the linear empathy tool]).

CONTACTS AND LOCATIONS:
Overall Officials: Kumar Alagappan, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M.D. Anderson Cancer Center — http://www.mdanderson.org